CLINICAL TRIAL: NCT03324230
Title: Exacerbation Profile in Patients on Mepolizumab for Severe Refractory Eosinophilic Asthma- an Exploratory Study.
Brief Title: Exploring Asthma Exacerbations in Mepolizumab Treated Patients
Status: Completed | Type: Observational
Sponsor: Queen's University, Belfast (Other)
Collaborators: RASP (Refractory Asthma Stratification Programme) (Unknown); Medical Research Council (Other Government); University of Oxford (Other); University of Leicester (Other); NHS Greater Glasgow and Clyde (Other); Belfast Health and Social Care Trust (Other)
Responsible Party: Principal Investigator, Liam Heaney, Professor, Queen's University, Belfast
Other Study IDs: B17/30
Record Dates: First submitted 2017-09-26; First posted 2017-10-27 (Actual); Last update posted 2019-07-10 (Actual); Status verified 2019-07

CONDITIONS: Asthma Brittle
Keywords: Monoclonal antibody; Mepolizumab; Eosinophil

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Whole blood, sputum, urine.
Oversight: FDA-regulated Device: No

SUMMARY:
This is a multicentre, observational study focusing on exacerbation events in patients with severe eosinophilic asthma on Mepolizumab.

Mepolizumab is an anti-IL5 (Interleukin 5) monoclonal antibody which blocks the eosinophilic activation pathways associated with decreasing asthma control. The pre-licensing studies have shown that Mepolizumab decreases asthma exacerbation events by approximately 50%, this study seeks to understand the underlying mechanisms of the remaining 50% of exacerbations.

The study will enrol patients within GINA classification 4 and 5 who are known to difficult asthma services across four UK sites. Some patients will recently have been commenced on Mepolizumab, whilst others will be commenced on the drug on entry to the study. The patients will have baseline measurements of biomarkers, lung function, sputum analysis and quality of life questionnaires on study entry, after which patients will be asked to contact the clinic at the first signs of worsening asthma symptoms to arrange a clinic visit prior to commencing rescue treatment. They will be clinically assessed with review of peak flow and symptom diaries, measurements taken at baseline will be repeated and a decision on the nature of the exacerbation and treatment required will be made.

This is an observational study, all outcomes will be exploratory.

DETAILED DESCRIPTION:
Background:

Around 15% of the United Kingdom (UK) have asthma, of these, 10-20% have asthma which is difficult to control using current therapies and with high levels of morbidity resulting. These patients consume 50-60% of the UK healthcare costs of asthma and as such, there is much interest in developing novel treatments for this group.

The heterogeneity of inflammatory pathways underlying asthma are of great interest with development of biomarkers useful for phenotyping asthmatic patients and allowing more accurate assessment of their response to treatment. Traditionally, oral corticosteroids are used in eosinophilic 'T2-high' asthmatic patients with good therapeutic effect, however, there are a group of T2-high patients who have refractory type-2 cytokine driven inflammation and airway eosinophilia despite oral corticosteroids. As such, there are several novel biological agents being engineered to block type 2 cytokine pathways including antagonists to IL5, IL13 and IL4 (Interleukin 5, 13, 4).

Mepolizumab is a humanised monoclonal antibody against IL5. Through a selective inhibition of eosinophilic inflammation, the agent reduces the number of eosinophils in sputum and blood, with important clinical outcomes such as a reduction of asthma exacerbations and a need for systemic glucocorticoids. The pre-licencing clinical trials have shown that selective inhibition of IL5 and presumptive removal of eosinophils reduces exacerbations by 50%, but while this is a significant reduction, patients with severe asthma continue to have severe exacerbations requiring systemic corticosteroid administration.

Therefore, the point of interest is eliciting the inflammatory phenotype and physiological characteristics of the remaining 50% of exacerbations and ascertaining whether systemic corticosteroids have a role when the IL-5 pathway has been blocked by Mepolizumab.

Purpose/ Aim This is an observational study designed to phenotype exacerbations or worsening asthma control when participants are established on Mepolizumab. The study will look for changes in lung function, biomarkers and patient symptoms scores.

The hypothesis is as follows: In patients with severe refractory eosinophilic asthma, who have been established on mepolizumab:

- increased asthma symptoms (exacerbations) will have no evidence of airway eosinophilia and will be clinically mild events associated with small reductions in lung function which may not require rescue oral corticosteroids.

Outline plan of investigation This will be an open observational multi-centre, cohort study in participants with severe asthma (Global Initiative for Asthma (GINA) Steps 4 and 5 classification of asthma severity) who are initiated on Mepolizumab in line with the NICE/SMC (National institute foe Health and Care Excellence) Clinical Guidelines.

The study is exploratory and will assess deteriorations in asthma control to characterise the clinical severity of each exacerbation and the airway and systemic inflammatory phenotype associated with these events. Clinical assessment and management of each exacerbation will be in line with standard clinical guidelines (SIGN 153 (Scottish Intercollegiate Guidelines Network), British Guideline on the Management of Asthma, September 2016).

The study design incorporates a proportion of participants already established on Mepolizumab as well as participants who will be commenced on Mepolizumab on entry to the study. A baseline assessment of medical history, clinical examination, lung function and sputum/blood/urine for analysis will be undertaken along with quality of life questionnaires. Those newly started on Mepolizumab, will be assessed in a similar manner 3 months into the study.

Subjects will be given an electronic peak flow recorder, symptoms diary and action plan for change in baseline symptoms. Participants will be asked to contact the clinic when they feel there has been a decline in asthma control and before they take rescue treatment, a clinic visit will be arranged. At this visit, all participants will have full medical assessment and clinical management based on detailed medical history, clinical findings and lung function measurement. Blood will be taken as part of this clinical assessment as outlined in the schedule of study procedures including biobanking of samples for whole blood gene expression, serum, plasma, sputum and urine. These samples will be stored for validation of additional biomarkers, aligned with the RASP-UK (Refractory Asthma Stratification Programme-UK) biomarker corticosteroid optimisation study.

Number in study:

This is a study will take place across 4 NHS sites within the UK, namely Belfast, Glasgow, Oxford and Leicester.

The study design incorporates a proportion of participants already established on Mepolizumab and also participants starting on Mepolizumab, allowing recruitment of up to 150 participants in a 6 - 9 month window (all sites have large numbers of patients on the waiting list for the drug). Assuming a conservative 0.7 exacerbations per patient per year on mepolizumab (ca 160 events in an 18 month period) and a minimum rate of attendance of 65% this is 102 observed episodes. The study will be terminated when 100 clinical assessments at exacerbation in total have been completed across all sites for participants on Mepolizumab prior to initiation of rescue treatment. The expected duration of study per participant is 24 months.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and ≤ 80 years at Visit 1
2. Able and willing to provide written informed consent and to comply with the study protocol including being able to contact the clinical center and to attend for assessment during a symptomatic deterioration
3. Severe asthma despite confirmed after assessment by an asthma specialist
4. Diagnosed with asthma at least 12 months prior to screening

Exclusion Criteria:

1. Acute exacerbation requiring oral corticosteroids in 4 weeks before screening.
2. Other clinically significant medical disease or uncontrolled concomitant disease despite treatment that is likely, in the opinion of the investigator, to require a change in therapy or impact the ability to participate in the study
3. History of current alcohol, drug, or chemical abuse or past abuse that would impair or risk the subject's full participation in the study, in the opinion of the investigator
4. Treatment with an investigational agent within 30 days of visit 1 (or 5 half-lives of the investigational agent, whichever is longer)
5. Female subjects who are pregnant or lactating (excluded as candidates for Mepolizumab in clinic prior to study)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients known to Difficult Asthma services within the NHS, who are eligible for Mepolizumab treatment as per NICE guidelines.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-29 (Actual); Study Completion 2019-06-29 (Actual)

PRIMARY OUTCOMES:
Number of asthma exacerbations requiring administration of corticosteroids | Throughout study completion, an average of 2 years
  Mepolizumab is considered to be a steroid sparing drug resulting in a reduced number of asthma exacerbations. Patients will be reviewed when asthma symptoms worsen to assess the cause of loss of asthma control and ascertain if the exacerbations requires administration of corticosteroids.
Forced Expiratory Volume in 1 second | Throughout study completion, an average of 2 years
  Spirometry to assess Forced Expiratory Volume in 1 (FEV1) second will be performed at baseline entry to the study and on worsening of asthma symptoms. Spirometry will performed in keeping with the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines.
Forced vital capacity | Throughout study completion, an average of 2 years
  Spirometry to assess Forced Vital Capacity (FVC) will be undertaken at baseline and at worsening of asthma symptoms. Spirometry will performed in keeping with the American Thoracic Society (ATS) and European Respiratory Society (ERS) guidelines.
Fractional expired nitric oxide (feno) | Throughout study completion, an average of 2 years
  Feno will be measured at baseline and during unscheduled visits to assess airway inflammation.
Mini-AQLQ | Throughout study completion, an average of 2 years
  The mini-Asthma Quality of Life Questionnaire (mini-AQLQ) will be used throughout the study to assess effect of asthma on the subject's quality of life.
Asthma control questionnaire (ACQ) | Throughout study completion, an average of 2 years
  The Asthma control questionnaire (ACQ) will be used throughout the study to assess effect of asthma on the subject's quality of life.
Saint George's Respiratory Questionnaire (SGRQ). | Throughout study completion, an average of 2 years
  The Saint George's Respiratory Questionnaire (SGRQ)will be used throughout the study to assess effect of asthma on the subject's quality of life.
Eosinophils | Throughout study completion, an average of 2 years
  Complete blood count with breakdown of individual cell counts will be measured at baseline and worsening of asthma symptoms
C reactive protein | Throughout study completion, an average of 2 years
  Serum C reactive protein will be measured at baseline and worsening of asthma symptoms.
Sputum analysis | Throughout study completion, an average of 2 years
  The breakdown of the sputum white cell count will be analysed to assess for eosinophilia and neutrophilia.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Heaney, MB Bch BaO, Principal Investigator — Queen's University, Belfast
Locations (4):
- United Kingdom (4):
  - Queen's University Belfast, Belfast, County Antrim
  - Leicester Biomedical Research Centre, Leicester, Leicestershire
  - Gartnavel General Hospital, Greater Glasgow and Clyde NHS Trust, Glasgow, Scotland
  - Oxford University, Oxford

REFERENCES:
- [Background] Smith DH, Malone DC, Lawson KA, Okamoto LJ, Battista C, Saunders WB. A national estimate of the economic costs of asthma. Am J Respir Crit Care Med. 1997 Sep;156(3 Pt 1):787-93. doi: 10.1164/ajrccm.156.3.9611072. PMID 9309994
- [Background] Barnes PJ, Jonsson B, Klim JB. The costs of asthma. Eur Respir J. 1996 Apr;9(4):636-42. doi: 10.1183/09031936.96.09040636. PMID 8726924
- [Background] Sweeney J, Brightling CE, Menzies-Gow A, Niven R, Patterson CC, Heaney LG; British Thoracic Society Difficult Asthma Network. Clinical management and outcome of refractory asthma in the UK from the British Thoracic Society Difficult Asthma Registry. Thorax. 2012 Aug;67(8):754-6. doi: 10.1136/thoraxjnl-2012-201869. Epub 2012 May 11. PMID 22581823
- [Background] Ahmad F, Roman J. Treating refractory asthma with antibodies against IL-5: is it ready for prime time? Expert Rev Respir Med. 2009 Jun;3(3):227-30. doi: 10.1586/ers.09.22. PMID 20477317
- [Background] Pavord ID, Korn S, Howarth P, Bleecker ER, Buhl R, Keene ON, Ortega H, Chanez P. Mepolizumab for severe eosinophilic asthma (DREAM): a multicentre, double-blind, placebo-controlled trial. Lancet. 2012 Aug 18;380(9842):651-9. doi: 10.1016/S0140-6736(12)60988-X. PMID 22901886
- [Background] Quanjer PH, Stanojevic S, Cole TJ, Baur X, Hall GL, Culver BH, Enright PL, Hankinson JL, Ip MS, Zheng J, Stocks J; ERS Global Lung Function Initiative. Multi-ethnic reference values for spirometry for the 3-95-yr age range: the global lung function 2012 equations. Eur Respir J. 2012 Dec;40(6):1324-43. doi: 10.1183/09031936.00080312. Epub 2012 Jun 27. PMID 22743675
- [Derived] McDowell PJ, Diver S, Yang F, Borg C, Busby J, Brown V, Shrimanker R, Cox C, Brightling CE, Chaudhuri R, Pavord ID, Heaney LG; Medical Research Council: Refractory Asthma Stratification Programme (RASP-UK Consortium). The inflammatory profile of exacerbations in patients with severe refractory eosinophilic asthma receiving mepolizumab (the MEX study): a prospective observational study. Lancet Respir Med. 2021 Oct;9(10):1174-1184. doi: 10.1016/S2213-2600(21)00004-7. Epub 2021 May 7. PMID 33971168
- See also: 2017 GINA Report, Global Strategy for Asthma Management and Prevention — http://ginasthma.org/2017-gina-report-global-strategy-for-asthma-management-and-prevention/